CLINICAL TRIAL: NCT04717752
Title: A Randomized Controlled Study of Different Trigger Modes of Antagonist Regimen in Patients With Low Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Reproductive Medicine Center, Drum Tower Hospital Affiliated to Nanjing University Medical College, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ-POR-DTMAR-2020
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Poor Ovarian Response
Keywords: poor ovarian response
MeSH Terms: interventions — Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double trigger unit (Experimental): HCG: 6000IU (Ovidrel: 250ug) + GnRH-a (Troprilin) 0.2mg
  Interventions: Drug: Ovidrel; Drug: Troprilin
- HCG trigger unit (Sham Comparator): HCG: 6000IU (Ovidrel: 250ug)
  Interventions: Drug: Ovidrel

INTERVENTIONS:
Drug: Ovidrel — recombinant human chorionic gonadotropin for injection
Drug: Troprilin — triptorelin acetate injection
  Arms: Double trigger unit

SUMMARY:
Assisted reproductive technology (ART), especially controlled ovarian stimulation (COS), significantly increased clinical pregnancy rates among infertile patients. However, about 9% to 24% of patients had poor ovarian response to gonadotropins (GNS) stimulation, which was called poor ovarian response (POR). In recent years, the diagnosis and treatment of patients with low fertility is the challenge for reproductive medicine. To better demonstrate the effectiveness of various interventions and distinguish the different subgroups of patients, 2016 POSEIDON (Patient-Oriented Strategies Encompassing Individualized Oocyte Number) standard changed low reaction into low prognosis of patient-oriented individual strategies to obtain eggs. For patients in group 3 and group 4 classified by POSEIDON, ovarian reserve function decline, follicular development desynchrony and low numbers of oocytes obtained lead to poor prognosis. In 2020, the prognosis based on Delphi method of assisted reproductive technology to treat low crowd diagnosis expert opinion in China recommended to give these patients conventional cosine solutions such as antagonist. In the first cycle, follicle stimulating hormone (FSH) starting dose of 225 ~ 300 iu is suggested to achieve plenty of ovarian stimulation for standards and maximize the benefits of superovulation. Because of the particularity of luteal support in the antagonist regimen, it is of great clinical significance to explore the trigger mode and combination mode of luteal support in the antagonist regimen for patients with poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 42 years old, AFC<5 and or AMH<1.2ng/ml ② Adopt antagonist program for controlled ovulation hyperstimulation (COH); patients with fresh cycle transplantation;

  * Accept conventional IVF or intracytoplasmic sperm injection (ICSI);

    * The ART treatment cycle is less than 3 times.

Exclusion Criteria:

* Abnormal chromosome karyotype;

  * Severe endometriosis;

    * Abnormal thyroid function; ④ Pregnancy contraindications; ⑤ Past history of ovarian tumors or after receiving radiotherapy

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate in each transplantation cycle | 6 weeks
  number of pregnant cases are confirmed by ultrasound/ total number of transplanted

SECONDARY OUTCOMES:
Rate of cancelled cycle | 6 weeks
  number of cancelled cycles/ number of total cycles
Number of mature eggs | 6 weeks
  number of matured oocytes
Number of high-quality embryos | 6 weeks
  number of D3 high quality embryos (≥7 scores)
Implantation rate | 6 weeks
  number of gestational sacs/ number of transplanted embryos
Early abortion rate | 6 weeks
  number of miscarriage cases/ number of pregnant cases confirmed by ultrasound
Cumulative pregnancy rate per stimulation cycle | 6 weeks
  number of pregnant cases which are confirmed by ultrasound/ total number of stimulation cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] Orvieto R. Triggering final follicular maturation--hCG, GnRH-agonist or both, when and to whom? J Ovarian Res. 2015 Aug 21;8:60. doi: 10.1186/s13048-015-0187-6. PMID 26293447
- [Background] Nakano R, Mizuno T, Kotsuji F, Katayama K, Wshio M, Tojo S. "Triggering" of ovulation after infusion of synthetic luteinizing hormone releasing factor (LRF). Acta Obstet Gynecol Scand. 1973;52(3):269-72. doi: 10.3109/00016347309158325. No abstract available. PMID 4582787
- [Background] Gonen Y, Balakier H, Powell W, Casper RF. Use of gonadotropin-releasing hormone agonist to trigger follicular maturation for in vitro fertilization. J Clin Endocrinol Metab. 1990 Oct;71(4):918-22. doi: 10.1210/jcem-71-4-918. PMID 2119392
- [Background] Griesinger G, Diedrich K, Devroey P, Kolibianakis EM. GnRH agonist for triggering final oocyte maturation in the GnRH antagonist ovarian hyperstimulation protocol: a systematic review and meta-analysis. Hum Reprod Update. 2006 Mar-Apr;12(2):159-68. doi: 10.1093/humupd/dmi045. Epub 2005 Oct 27. PMID 16254001
- [Background] Griesinger G, Kolibianakis EM, Papanikolaou EG, Diedrich K, Van Steirteghem A, Devroey P, Ejdrup Bredkjaer H, Humaidan P. Triggering of final oocyte maturation with gonadotropin-releasing hormone agonist or human chorionic gonadotropin. Live birth after frozen-thawed embryo replacement cycles. Fertil Steril. 2007 Sep;88(3):616-21. doi: 10.1016/j.fertnstert.2006.12.006. Epub 2007 Apr 23. PMID 17451691
- [Background] Youssef MA, Van der Veen F, Al-Inany HG, Mochtar MH, Griesinger G, Nagi Mohesen M, Aboulfoutouh I, van Wely M. Gonadotropin-releasing hormone agonist versus HCG for oocyte triggering in antagonist-assisted reproductive technology. Cochrane Database Syst Rev. 2014 Oct 31;2014(10):CD008046. doi: 10.1002/14651858.CD008046.pub4. PMID 25358904
- [Background] Griesinger G, Meldrum D. Introduction: Management of the luteal phase in assisted reproductive technology. Fertil Steril. 2018 May;109(5):747-748. doi: 10.1016/j.fertnstert.2018.02.009. PMID 29778366
- [Background] Lawrenz B, Coughlan C, Fatemi HM. Individualized luteal phase support. Curr Opin Obstet Gynecol. 2019 Jun;31(3):177-182. doi: 10.1097/GCO.0000000000000530. PMID 30855289
- [Background] Griffin D, Benadiva C, Kummer N, Budinetz T, Nulsen J, Engmann L. Dual trigger of oocyte maturation with gonadotropin-releasing hormone agonist and low-dose human chorionic gonadotropin to optimize live birth rates in high responders. Fertil Steril. 2012 Jun;97(6):1316-20. doi: 10.1016/j.fertnstert.2012.03.015. Epub 2012 Apr 3. PMID 22480822
- [Background] Schachter M, Friedler S, Ron-El R, Zimmerman AL, Strassburger D, Bern O, Raziel A. Can pregnancy rate be improved in gonadotropin-releasing hormone (GnRH) antagonist cycles by administering GnRH agonist before oocyte retrieval? A prospective, randomized study. Fertil Steril. 2008 Oct;90(4):1087-93. doi: 10.1016/j.fertnstert.2007.07.1316. Epub 2007 Nov 26. PMID 18023439
- [Background] Li S, Zhou D, Yin T, Xu W, Xie Q, Cheng D, Yang J. Dual trigger of triptorelin and HCG optimizes clinical outcome for high ovarian responder in GnRH-antagonist protocols. Oncotarget. 2018 Jan 4;9(4):5337-5343. doi: 10.18632/oncotarget.23916. eCollection 2018 Jan 12. PMID 29435182
- [Background] Eftekhar M, Mojtahedi MF, Miraj S, Omid M. Final follicular maturation by administration of GnRH agonist plus HCG versus HCG in normal responders in ART cycles: An RCT. Int J Reprod Biomed. 2017 Jul;15(7):429-434. PMID 29177244
- [Background] Lin MH, Wu FS, Lee RK, Li SH, Lin SY, Hwu YM. Dual trigger with combination of gonadotropin-releasing hormone agonist and human chorionic gonadotropin significantly improves the live-birth rate for normal responders in GnRH-antagonist cycles. Fertil Steril. 2013 Nov;100(5):1296-302. doi: 10.1016/j.fertnstert.2013.07.1976. Epub 2013 Aug 28. PMID 23993928
- [Background] Zhou X, Guo P, Chen X, Ye D, Liu Y, Chen S. Comparison of dual trigger with combination GnRH agonist and hCG versus hCG alone trigger of oocyte maturation for normal ovarian responders. Int J Gynaecol Obstet. 2018 Jun;141(3):327-331. doi: 10.1002/ijgo.12457. Epub 2018 Feb 21. PMID 29388691
- [Background] Lu X, Hong Q, Sun L, Chen Q, Fu Y, Ai A, Lyu Q, Kuang Y. Dual trigger for final oocyte maturation improves the oocyte retrieval rate of suboptimal responders to gonadotropin-releasing hormone agonist. Fertil Steril. 2016 Nov;106(6):1356-1362. doi: 10.1016/j.fertnstert.2016.07.1068. Epub 2016 Aug 1. PMID 27490046
- [Background] Griffin D, Feinn R, Engmann L, Nulsen J, Budinetz T, Benadiva C. Dual trigger with gonadotropin-releasing hormone agonist and standard dose human chorionic gonadotropin to improve oocyte maturity rates. Fertil Steril. 2014 Aug;102(2):405-9. doi: 10.1016/j.fertnstert.2014.04.028. Epub 2014 May 17. PMID 24842671
- [Background] Gold JI, Stocker AA. Visual Decision-Making in an Uncertain and Dynamic World. Annu Rev Vis Sci. 2017 Sep 15;3:227-250. doi: 10.1146/annurev-vision-111815-114511. Epub 2017 Jul 17. PMID 28715956
- [Background] Belova EV, Emtseva VP, Obolenskii IuA. [Characteristics of autonomic and hormonal reactions during the performance of different types of intellectual work]. Fiziol Cheloveka. 1988 May-Jun;14(3):482-5. No abstract available. Russian. PMID 2844614
- [Background] Deepika K, Rathore S, Garg N, Rao K. Empty follicle syndrome: Successful pregnancy following dual trigger. J Hum Reprod Sci. 2015 Jul-Sep;8(3):170-4. doi: 10.4103/0974-1208.165152. PMID 26538861
- [Background] Zilberberg E, Haas J, Dar S, Kedem A, Machtinger R, Orvieto R. Co-administration of GnRH-agonist and hCG, for final oocyte maturation (double trigger), in patients with low proportion of mature oocytes. Gynecol Endocrinol. 2015 Feb;31(2):145-7. doi: 10.3109/09513590.2014.978850. Epub 2014 Nov 11. PMID 25385007
- [Background] Oliveira SA, Calsavara VF, Cortes GC. Final Oocyte Maturation in Assisted Reproduction with Human Chorionic Gonadotropin and Gonadotropin-releasing Hormone agonist (Dual Trigger). JBRA Assist Reprod. 2016 Dec 1;20(4):246-250. doi: 10.5935/1518-0557.20160047. PMID 28050961
- [Background] Eser A, Devranoglu B, Bostanci Ergen E, Yayla Abide C. Dual trigger with gonadotropin-releasing hormone and human chorionic gonadotropin for poor responders. J Turk Ger Gynecol Assoc. 2018 Jun 4;19(2):98-103. doi: 10.4274/jtgga.2017.0045. Epub 2018 Mar 8. PMID 29516855
- [Background] Lin MH, Wu FS, Hwu YM, Lee RK, Li RS, Li SH. Dual trigger with gonadotropin releasing hormone agonist and human chorionic gonadotropin significantly improves live birth rate for women with diminished ovarian reserve. Reprod Biol Endocrinol. 2019 Jan 4;17(1):7. doi: 10.1186/s12958-018-0451-x. PMID 30609935
- [Background] Ding N, Liu X, Jian Q, Liang Z, Wang F. Dual trigger of final oocyte maturation with a combination of GnRH agonist and hCG versus a hCG alone trigger in GnRH antagonist cycle for in vitro fertilization: A Systematic Review and Meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Nov;218:92-98. doi: 10.1016/j.ejogrb.2017.09.004. Epub 2017 Sep 14. PMID 28957685